CLINICAL TRIAL: NCT02342054
Title: Prospective Phase II Trial of Single Fraction Real-time High-Dose-Rate (19-HDR) Brachytherapy in Patients With Low and Intermediate Risk Prostate Cancer
Brief Title: Single Fraction Real-time High-Dose-Rate Brachytherapy in Patients With Low and Intermediate Risk Prostate Cancer
Acronym: SINFRA_PROST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Cruces (Other)
Responsible Party: Principal Investigator, Alfonso Gomez-Iturriaga, Staff physician department of Radiation Oncology, Hospital de Cruces
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINFRA_PROST
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
Keywords: Cancer; Prostate Cancer; Brachytherapy; Dose escalation; High Dose Rate; MRI-TRUS fusion; Detection of DILs by MRI; SINGLE FRACTION
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI-TRUS fusion guided Single Frac HDR (Experimental): Patients treated with a Single Fraction Real-Time High-Dose-Rate (HDR 19Gy)
  Interventions: Radiation: MRI-TRUS fusion guided Single Frac HDR

INTERVENTIONS:
Radiation: MRI-TRUS fusion guided Single Frac HDR
  Other Names: Single Fraction real time HDR (19Gy); Planning software Oncentra Prostate for Nucletron

SUMMARY:
High-dose rate brachytherapy (HDR-BT) is an advanced technology theorized to be more advantageous than LDR-BT and External Beam Radiotherapy (EBRT), to the patient himself, and in terms of resource allocation. Studies of HDR-BT monotherapy have encouraging results in terms of biochemical control, patient survival and toxicity, but there are still certain limitations that preclude recommending HDR-BT monotherapy outside the setting of a clinical trial.

The primary endpoint of this study is to evaluate the safety, tolerance and impact on quality of life (QoL) of the BT-HDR 19Gy administered in single fraction in patients with low and intermediate risk prostate cancer. Secondary endpoint is to measure the efficacy, in terms of cancer control and satisfaction of the patients undergoing the experimental treatment.

Forty nine patients will be recruited for the experimental procedure Quality of Life, tolerance, gastrointestinal and genitourinary toxicity will be assessed using standardized procedures and scales. Patient satisfaction with the procedure will be appraised using five-category predetermined Likert scale questions.

Two different types of intermediate analyses will be performed: with 15 and 30 recruited patients.

The experimental treatment tested in this study is very innovative. Since prostate cancer is the most frequent cancer in men in Spain, this trial results are very likely to have a major impact on the standard therapy for prostate cancer in our National Health Service, allowing for a higher number of Hospitals within our country and other countries starting protocols of HDR BT 19Gy in single fraction.

DETAILED DESCRIPTION:
Treatment:

The patient´s treatment will consist of MRI-TRUS fusion single HDR brachytherapy fraction (1 fraction of 1900 cGray).

Brachytherapy performed under general anesthesia as an outpatient procedure

TRUS-MRI fusion:

T2 axial volumetric sequence (VISTA) is imported directly from the picture archiving and communication systems (PACS). Then MR images are reconstructed and segmented. Target volumes (prostate gland, dominant intraprostatic lesions (DILs) Organs at risk (OARs) urethra and rectum are delineated.

A transrectal sagittal volumetric ultrasound image is immediately acquired every 2 degrees, a rapid reconstruction algorithm converts the series of 2D images into a 3D volume, which is then displayed in axial, sagittal and coronal views and transferred to the module of fusion with the MRI.

The MRI images and the real-time sonography examination are displayed on a split-screen with the possibility of overlaying the images live in one image. A graphical user interface is used for rigid manual registration of the ultrasound and MRI volumes. This interface allows for displacements in the three dimensions and rotations, until both images are correctly superimposed.

Then the contoured structures are transferred to the US dataset, and these contours are slightly modified until a perfect matching with the US images is achieved.

Dose prescription:

Ultrasound images with the catheters in place will be exported to Oncentra Prostate. The prostate, Foley catheter and anterior rectal wall will be contoured. Catheters will be reconstructed on the planning system. Anatomy based inverse planning will be used for dwell time optimization.

The homogeneity parameters used for optimization aim are:

-For prostate V100 > 95%, V150 <35%, V200 < 6%, where Vn is the fractional volume of the organ that receives n% of the prescribed dose.

The dose constraints for the organ at risk will be:

* Urethral dmax < 110% and
* Rectal 1cc < 60% of prescribed dose.

Endpoints

Feasibility of higher doses administration, toxicity and efficacy will be measured

ELIGIBILITY:
Inclusion Criteria:

* Men older than 18 years old
* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Clinical stage T1c/T2a disease
* Low and Intermediate risk disease defined as either Gleason 6 or Gleason 7 and PSA < 20 ng/ml.
* Prostate volume < 60 cc as determined by ultrasound, CT or MRI
* Life expectancy of more than 10 years
* Willing to give informed consent to participate in this clinical trial
* Able and willing to complete Expanded Prostate Index Composite (EPIC) questionnaire
* Eastern Cooperative Oncology Group (ECOG) of 0 - 2.
* Give competent informed consent to participate in this trial.

Exclusion Criteria:

* Documented nodal or distant metastases
* Previous pelvic radiotherapy
* Previous trans-urethral resection of prostate, previous prostatectomy or HIFU
* Use of androgen deprivation therapy. Use of 5-alpha-reductase inhibitors is permitted
* Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >19
* Contra-indication to radical prostate radiotherapy
* Significant medical co-morbidity rendering patient unsuitable for general anaesthetic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety measured by i) urinary retention rate and duration ii) maximum International Prostate Symptom Score and time to normalize | 12 months
  Data to be collected are:
  i) urinary retention rate and duration ii) maximum International Prostate Symptom Score and time to normalize
Quality of Life measured by alidated instruments including International Prostate Symptom Score and the urinary, bowel and sexual domains of EPIC | 12 months
  Quality of life will be measured through validated instruments including International Prostate Symptom Score and the urinary, bowel and sexual domains of EPIC

SECONDARY OUTCOMES:
Acute toxicity measured by urinary retention rate, International Prostate Symptom Score over time, rectal toxicity and genitourinary toxicity | 24 months
  Data to be collected: urinary retention rate, International Prostate Symptom Score over time, rectal toxicity and genitourinary toxicity
Efficacy, measured by PSA | 24 months
  Patients will be followed with PSA at every follow-up;
Patient satisfaction measured with Likert scale question | 24 months
  Patient Satisfaction will be measured with Likert scale question

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Gomez-Iturriaga, MD, PhD, Principal Investigator — Hospital Universitario Cruces/Biocruces
Locations (1):
- Hospital Universitario Cruces, Barakaldo, Bizkaia, Spain

REFERENCES:
- [Derived] Gomez-Iturriaga A, Casquero F, Pijoan JI, Minguez P, Espinosa JM, Irasarri A, Bueso A, Cacicedo J, Buchser D, Bilbao P. Health-related-quality-of-life and toxicity after single fraction 19 Gy high-dose-rate prostate brachytherapy: Phase II trial. Radiother Oncol. 2018 Feb;126(2):278-282. doi: 10.1016/j.radonc.2017.10.039. Epub 2017 Nov 15. PMID 29153462